CLINICAL TRIAL: NCT03260088
Title: Evaluation Of Pleural Effusion At Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nermen Abuelkassem, Dr, Assiut University
Other Study IDs: PLEFF
Record Dates: First submitted 2017-08-17; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with pleural effusion: In patients with pleural effusion that remains undiagnosed with common diagnostic algorithm, immunoglobulin G4 will be done in pleural fluid
  Interventions: Diagnostic Test: Immunoglobulin G4

INTERVENTIONS:
Diagnostic Test: Immunoglobulin G4 — IgG4 will be purified from pleural fluids by diethylaminoethyl (DEAE)-cellulose ion exchange nephlometry

SUMMARY:
Pleural effusion is an accumulation of fluid between the tissue layers that line the lungs and chest cavity. It has an estimated prevalence of 320 per 100,000 people in industrialized countries. The cause of the pleural effusion remains unclear in a substantial percentage of patients with persistently exudative effusions.

DETAILED DESCRIPTION:
They are classified broadly into exudative and transudative effusion based on Light's criteria.

Several methods have been proposed for the identification of pleural effusion etiology including pleural fluid cytology, pleural biopsy, thoracoscopy and computerized tomography. However, these technologies have their own limitations.

The diagnosis of malignant pleural effusion is a vexing problem, since pleural fluid cytology findings are positive in only 60% of cases on average. Tumor marker carcinoembryonic antigen (CEA) can be positive in 80% of cases.

Thoracoscopy will establish the diagnosis in approximately 95% of cases, but this interventional procedure may not be available at all facilities.

A new approach is needed to detect the cause of undiagnosed pleural effusions. Diagnosis of idiopathic pleural effusion was made after a minimum of one year follow up with detailed exploration including computed tomographic scanning to exclude other causes of effusion such as malignant pleural effusion.

Because immunoglobulin G4 (IgG4)-related disease is recognized as a fibroinflammatory condition of unknown cause that can affect multiple organs including the lungs and pleura, IgG4 might be related to certain idiopathic pleural effusions.

The criteria of Common radiological findings of IgG4-related lung disease include hilar and mediastinal lymphadenopathy, thickening of perilymphatic interstitium with or without subpleural and/or peribronchovascular consolidation.

ELIGIBILITY:
Inclusion Criteria:

* All patients with exudative pleural effusion admitted to Assiut university hospital in period of October 2017 to October 2018

Exclusion Criteria:

* Patients with transudative pleural effusion

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with exudative pleural effusion admitted to Assiut university hospital in period of October 2017 to October 2018
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2017-10-30 (Estimated); Primary Completion 2019-10-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
diagnosis new causes of previously remained undiagnosed cases of pleural effusion by using IgG4 in Assiut university hospital | one year
  Immunoglobulin G4 will be puified from pleural fluids by diethylaminoetyyl cellulose ion exchange nephlometry in patients with undiagnosed effusion after common investigations as it positive in IgG4 related disease. The median effusion IgG4 level was 41mg/dl in the IgG4 positive group and 27mg/dl in the IgG negative group.

CONTACTS AND LOCATIONS:
Overall Officials: Raafat T Elsokary, Prof, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Della-Torre E, Lanzillotta M, Doglioni C. Immunology of IgG4-related disease. Clin Exp Immunol. 2015 Aug;181(2):191-206. doi: 10.1111/cei.12641. Epub 2015 Jun 8. PMID 25865251
- [Background] Davies HE, Nicholson JE, Rahman NM, Wilkinson EM, Davies RJ, Lee YC. Outcome of patients with nonspecific pleuritis/fibrosis on thoracoscopic pleural biopsies. Eur J Cardiothorac Surg. 2010 Oct;38(4):472-7. doi: 10.1016/j.ejcts.2010.01.057. Epub 2010 Mar 12. PMID 20219385
- [Background] Ferrer JS, Munoz XG, Orriols RM, Light RW, Morell FB. Evolution of idiopathic pleural effusion: a prospective, long-term follow-up study. Chest. 1996 Jun;109(6):1508-13. doi: 10.1378/chest.109.6.1508. PMID 8769502